CLINICAL TRIAL: NCT02038660
Title: Evaluation of Effectiveness and Safety of Drug-Eluting Balloon in Routine Clinical Practice; A Multicenter Prospective Observational Cohort Study
Brief Title: Drug-Eluting Balloon Registry in Routine Clinical Practice
Acronym: IRIS DEB
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); B. Braun Korea Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2013-10
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Angioplasty, Balloon
Keywords: Coronary Artery Disease; Angioplasty, Balloon
MeSH Terms: conditions — Coronary Artery Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with coronary artery disease
  Interventions: Device: Balloon angioplasty

INTERVENTIONS:
Device: Balloon angioplasty

SUMMARY:
The purpose of this study is to evaluate long-term effectiveness and safety of patients with coronary disease treated with drug eluting balloon in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* After pre dilatation residual stenosis 30% and less and also without vessel dissection interrupted blood flow
* Age 20 and more
* Treated with Balloon angioplasty
* Signed informed consent and agreed to follow protocol

Exclusion Criteria:

* Allergy to paclitaxel, antiplatelet
* History of side effect to heparin, aspirin, thienopyridines
* History of bleeding tendency, coagulation disorder, blood transfusion reaction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with balloon angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Composite Event | 1year
  Death, Non-fatal myocardial infarction, Target vessel revascularization

SECONDARY OUTCOMES:
All cause death | 5year
Cardiac death | 5year
Myocardial infarction | 5year
Composite event | 5year
  Death or myocardial infarction
Composite event | 5year
  Cardiac death or myocardial infarction
Target vessel revascularization | 5year
Target lesion revascularization | 5year
Stent thrombosis | 5year
  Classification of stent thrombosis according to Academic Research Consortium criteria
Stroke | 5year
Procedural Success | 3day
  Defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization.
  Participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Dong-A Medical Center, Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.